CLINICAL TRIAL: NCT06524128
Title: PARA-DREEFT : Evaluation of Perceived Satisfaction With the Use of the Dreeft® Device in Real-life Situations
Brief Title: Evaluation of Perceived Satisfaction With the Use of the Dreeft® Device in Real-life Situations
Acronym: PARA-DREEFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles de Kerpape (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-A00781-46
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: People With Motor Disabilities

STUDY DESIGN:
Intervention Model Description: This is a randomized, bicentric, single-blind, cross-over study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With Dreeft® wheels (Experimental): The participant's wheelchair will be equipped with DREEFT wheels, to be used for 1 month.
  Interventions: Device: Dreeft wheels (EPPUR company)
- without Dreeft® wheels (No Intervention): The participant's wheelchair will be equipped with its usual braking system, monitored over a period of 1 month.

INTERVENTIONS:
Device: Dreeft wheels (EPPUR company) — The braking system (Dreeft wheels) is installed directly on the participant's wheelchair, by a trained occupational therapist. The Dreeft wheels are supplied for a period of 1 month.
  Arms: With Dreeft® wheels

SUMMARY:
Functional, independent mobility is essential for everyone (Fasciglione, 2017). It determines everyone's ability to engage in activities of daily living and contributes to maintaining health and well-being (Fasciglione, 2017).

However, the number of people with mobility limitations is increasing. Indeed, due to the aging of the population and the growing number of people with chronic diseases, the prevalence of people experiencing mobility-related limitations is increasing rapidly (Berardi et al., 2021); in addition to this health problems (such as osteoarticular, muscular, neurological diseases) and accidents are the cause of 23.6% and 42% of mobility-related limitation situations respectively (Camirand & Institut de la statistique du Québec, 2011).

To overcome these limitations, some people require the use of a manual wheelchair to enable mobility. Globally, wheelchair mobility (manual or motorized) refers to "the ability to move independently with a wheelchair, and to overcome obstacles encountered in carrying out activities of daily living or social roles" (Routhier et al., 2003, p. 20). This definition emphasizes that the use of a wheelchair enables independent movement.

In the past, the wheelchairs available were limited, expensive and rudimentary. Recent technological advances have given people access to a wide range of devices, adaptable to the majority of motor impairments and enabling movement in a wider variety of environments. Today's manual wheelchairs are increasingly sophisticated. However, they have no braking system other than the immobilizer that locks the wheels. Users have no choice but to use their hands as brake pads when gripping the handrail to slow down and stop.

A preliminary survey conducted by EPPUR among 164 manual wheelchair users, between March and May 2020, has shown that 75% of manual wheelchair users express difficulty braking with their wheelchair or resort to assistance from a third party (EPPUR). Worryingly, 50% of survey respondents reported having lost control of their wheelchair on a slope or ramp. Finally, in their daily lives, 85% of respondents reported having already changed their route to avoid a slope. For wheelchair users, negotiating sloping streets means constant braking.

The Dreeft® system was developed on the basis of these observations. No other system for braking manual wheelchairs is currently available. As described in the previous sections, the technology developed is based on the design of the hub which integrates the braking system, operating by back-pedaling. The manual wheelchair user benefits from improved responsiveness and manoeuvrability, with no friction on the hands. Adapted to manual wheelchairs, this innovative braking system is a potential revolution for users.

In order to confirm the benefits and functional contribution of the Dreeft® device in real life, a clinical study will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years and < to 64 years.
* Participants having signed the written consent form to participate in the study after free and informed information.
* Wheelchair user for more than one year.
* Participants affiliated to a social security scheme (beneficiary or beneficiary's beneficiary) excluding AME.
* Living at home.
* Have a motor disability, whatever its origin, and use a manual wheelchair independently as their main mobility tool, with or without propulsion assistance.
* Who propel their manual wheelchair with both upper limbs.
* Using a personal manual wheelchair compatible with Dreeft® wheels.
* Able to mount/dismount the wheels, or a third party to assist with wheel changes.
* Referred by the person's referring physician or occupational therapist on clinical indication for the device.

Exclusion Criteria:

* Participant deprived of liberty (by judicial or administrative decision).
* Participant of legal age under legal protection or unable to express consent.
* Participation in another ongoing clinical trial.
* Pregnant or breastfeeding women or women of childbearing age without contraception.
* Lack of proficiency in spoken and written French.
* Unstable health condition.
* Mentally or linguistically incapable of understanding the instructions for taking the research tests.
* User unable to propel himself/herself independently in a manual wheelchair, hemiplegic user.
* Body weight > 120 kg

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Canadian Measure of Occupational Performance (CMOP) - satisfaction score | 2 months
  The Canadian Measure of Occupational Performance (CMOP) will be used to assess changes in perceived satisfaction with daily living tasks identified as priorities by the user, and involving mobility with the wheelchair.

SECONDARY OUTCOMES:
Canadian Measure of Occupational Performance (CMOP) - performance score | 2 months
  The Canadian Measure of Occupational Performance (CMOP) will also be used to determine changes in perceived performance during the performance of daily living tasks identified as priorities by the user and involving a mobility action with the wheelchair.
F-PIADS scale | 2 months
  Evlaluaiton of the psychosocial impact of a technical aid (using the F-PIADS scale)
Wheelchair skill test - Questionnaire (WST-Q) | 2 months
  Evaluation of the manual wheelchair driving
QUEST measurement scale (Quebec User Evaluation of Satisfaction with assistive Technology) | 2 months
  Evaluation of satisfaction with a technical aid
Vancouver scale | 2 months
  Evaluation of changes in skin condition of hands Medical assessment
Number of people who would like to continue using the Dreeft® device and device abandonment rate | 2 months
  Questionnaires
Safety of use | 2 months
  Recording of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de rééducation et de réadaptation fonctionnelles de Kerpape, Ploemeur
  - Centre de ressources et d'innovation mobilité handicap (CEREMH), Vélizy-Villacoublay

IPD SHARING:
Plan to Share IPD: No